CLINICAL TRIAL: NCT01229228
Title: A Phase 2, Randomized, Double-Blind, Single-Dose, Parallel-Group, Active- and Placebo-Controlled Study of Naproxen [Test] Capsules for the Treatment of Pain After Surgical Removal of Impacted Third Molars
Brief Title: Study of Naproxen Capsules to Treat Dental Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Iroko Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NAP2-08-03
Record Dates: First submitted 2010-10-25; First posted 2010-10-27 (Estimated); Results first posted 2012-03-29 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-03

CONDITIONS: Dental Pain
MeSH Terms: conditions — Toothache | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Naproxen Test (lower dose) (Experimental): 200-mg
  Interventions: Drug: Naproxen Test
- Naproxen Test (upper dose) (Experimental): 400-mg (2 x 200-mg)
  Interventions: Drug: Naproxen Test
- Naprosyn 250 mg (Active Comparator)
  Interventions: Drug: Naprosyn
- Naprosyn 500 mg (Active Comparator)
  Interventions: Drug: Naprosyn
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naproxen Test — 200-mg single dose
  Arms: Naproxen Test (lower dose)
Drug: Naproxen Test — 400-mg (2 x 200-mg)
  Arms: Naproxen Test (upper dose)
Drug: Naprosyn — single dose
  Arms: Naprosyn 250 mg
Drug: Naprosyn — single dose
  Arms: Naprosyn 500 mg
Drug: Placebo — single dose
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether Naproxen Test Formulation Capsules are safe and effective for the treatment of dental pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female between 18 and 50 years of age
* For women of child-bearing potential: a woman who is not pregnant and not nursing, and who is practicing an acceptable method of birth control
* Patient requires extraction of 2 or more third molars
* Patient must be willing to stay at the study site overnight

Exclusion Criteria:

* Patient has hypersensitivity, allergy, or clinically significant intolerance to any medications to be used in the study, or related drugs
* Patient has a current disease or history of a disease that will impact the study or the patient's well-being
* Patient has used or intends to use any of the medications that are prohibited by the protocol
* Patient has a history of drug or alcohol abuse or dependence, or patient has a positive urine drug screen or alcohol breathalyzer test
* Patient has taken another investigational drug within 30 days prior to screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 254 (Actual)
Dates: Start 2010-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Premier Research Group Limited, Austin, Texas, United States

REFERENCES:
- [Derived] Young CL, Strand V, Altman R, Daniels S. A phase 2 study of naproxen submicron particle capsules in patients with post-surgical dental pain. Adv Ther. 2013 Oct;30(10):885-96. doi: 10.1007/s12325-013-0057-9. Epub 2013 Oct 15. PMID 24127200

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naproxen Test (Lower Dose) | Naproxen Test (Upper Dose) | Naprosyn 250 mg | Naprosyn 500 mg | Placebo
Started | 51 | 51 | 50 | 51 | 51
Completed | 50 | 51 | 49 | 51 | 50
Not Completed | 1 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naproxen Test (Lower Dose) | Naproxen Test (Upper Dose) | Naprosyn 250 mg | Naprosyn 500 mg | Placebo | Total
Number analyzed (Participants) | 51 | 51 | 50 | 51 | 51 | 254
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 51 | 51 | 50 | 51 | 51 | 254
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 21.1 (2.93) | 21.1 (3.29) | 20.7 (2.20) | 20.9 (2.88) | 21.1 (3.02) | 21.0 (2.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 30 | 32 | 21 | 32 | 148
  Male | 18 | 21 | 18 | 30 | 19 | 106
Region of Enrollment [Number; unit: participants]
  United States | 51 | 51 | 50 | 51 | 51 | 254

OUTCOME MEASURES:

1. Primary Outcome: Analysis of Total Pain Relief (TOTPAR) Over 0 to 12 Hours (TOTPAR-12) After Time 0
Description: Total pain relief as computed as a time-weighted sum of individual patient pain relief scores at each timepoint from 0-12 hours.
  Values for TOTPAR are measured from 0 to 4 on the Pain Relief Scale 0 None Min; 1 A little; 2 Some; 3 A lot; 4 Complete Max
  The TOTPAR is a weighted measure of the observations; the minimum possible value is 0 and the maximum possible value is 60.
Time Frame: Over 0 to 12 Hours
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Naproxen Test (Lower Dose): 200-mg single dose
Arm/Group | Naproxen Test (Lower Dose) | Naproxen Test (Upper Dose) | Naprosyn 250 mg | Naprosyn 500 mg | Placebo
Number analyzed (Participants) | 50 | 51 | 50 | 51 | 51
units on a scale | 25.868 [21.943 to 29.792] | 31.948 [28.065 to 35.831] | 24.373 [20.442 to 28.304] | 28.549 [24.660 to 32.439] | 9.531 [5.646 to 13.416]
Statistical Analysis 1: Comparison: Naproxen Test (Upper Dose) vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 22.417, 95% CI 2-sided [16.923 to 27.910], Standard Error of Mean 2.7891

ADVERSE EVENTS:
Arm/Group | Naproxen Test (Lower Dose) | Naproxen Test (Upper Dose) | Naprosyn 250 mg | Naprosyn 500 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/50 | 0/51 | 0/50 | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 28/51 | 27/51 | 25/50 | 26/51 | 31/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naproxen Test (Lower Dose) (N=50) | Naproxen Test (Upper Dose) (N=51) | Naprosyn 250 mg (N=50) | Naprosyn 500 mg (N=51) | Placebo (N=51)
Adverse drug reaction (General disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Naproxen Test (Lower Dose) (N=51) | Naproxen Test (Upper Dose) (N=51) | Naprosyn 250 mg (N=50) | Naprosyn 500 mg (N=51) | Placebo (N=51)
Dizziness (Nervous system disorders) | 5 | 3 | 2 | 0 | 6
Headache (Nervous system disorders) | 5 | 6 | 6 | 5 | 9
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 6 | 2 | 8 | 6 | 9
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 4 | 3 | 1 | 3
Post procedural swelling (Injury, poisoning and procedural complications) | 16 | 12 | 11 | 15 | 9
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No